CLINICAL TRIAL: NCT01118130
Title: Canadian Pharmacogenomics Network for Drug Safety: Genetic Factors Associated With Multiple Sclerosis Treatment
Brief Title: Pharmacogenomics of Drug Safety in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canada Foundation for Innovation (Other); Genome Canada (Other); British Columbia Clinical Genomics Network (Other)
Responsible Party: Principal Investigator, Bruce Carleton, Principle Investigator, University of British Columbia
Other Study IDs: H10-00494
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Genetics; genomics; Multiple Sclerosis; beta-interferons
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: MS patients experiencing an adverse drug reaction to an MS immunomodulatory therapy
- Control: MS patients not experiencing an adverse drug reaction to an MS immunomodulatory therapy

SUMMARY:
To investigate whether genotypic differences can be identified between MS patients developing 'liver injury' (defined as ALT levels five times the upper normal limit and above) compared to those not developing liver injury after exposure to beta-interferon for MS.

DETAILED DESCRIPTION:
PURPOSE: To investigate whether genotypic differences can be identified between MS patients who develop liver injury compared to those who do not develop injury in response to beta-interferon therapy.

OBJECTIVE: To determine whether elevated liver enzyme tests (ALT > 5 times the upper limit of normal) in response to beta-interferon therapy in MS patients is associated with genetic polymorphisms.

METHOD OF RECRUITMENT:

Patients will be identified through a clinic database and chart reviews. An introductory letter will be mailed to potential participants, inviting them to volunteer. A follow-up phone call will be made to determine interest and consent into study.

PROCEDURES:

Saliva will be collected for genetic analyses and a questionnaire will be administered

ELIGIBILITY:
Inclusion Criteria: Cases and controls must have

* definite MS (Poser or McDonald criteria)
* relapsing-remitting or secondary-progressive disease course
* Prescribed a beta-interferon as their immunomodulatory drug for MS

Exclusion Criteria:

* primary-progressive MS
* an elevated liver test result within 6 months of starting beta-interferon treatment
* presence of a co-morbidity that is a known risk-factor for liver injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple sclerosis (MS) patients attending MS clinics located at the University of British Columbia Hospital, Winnipeg Health Sciences Centre, Dalhousie (Halifax, Nova Scotia) MS clinic, London Health Sciences Centre (London, ON) and Hôpital Notre-Dame (Montréal). Participants must have definite MS (Poser or McDonald criteria), with a relapsing-remitting or secondary-progressive disease course, registered at one of the above MS Clinics and prescribed a beta-interferon as an immunomodulatory drug for MS.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-06 (Actual); Primary Completion 2025-05 (Actual); Study Completion 2025-05 (Actual)

PRIMARY OUTCOMES:
Experienced an adverse drug reaction or not? | No specified time frame

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Carleton, Principal Investigator — University of British Columbia; Michael Hayden, Study Director — University of British Columbia; Helen Tremlett, Study Director — University of British Columbia; Anthony Traboulsee, Study Director — University of British Columbia
Locations (5):
- Canada (5):
  - MS Clinic UBC Hospital, Vancouver, British Columbia
  - Winnipeg Health Sciences Centre, Winnipeg, Manitoba
  - Dalhousie MS Research Unit, Halifax, Nova Scotia
  - London Health Sciences Centre MS clinic, London, Ontario
  - Hôpital Notre-Dame MS clinic, Montreal, Quebec